CLINICAL TRIAL: NCT04428229
Title: The Evaluation of Optic Nerve Sheath Diameter in Patients Underwent Laparoscopic Colon and Gynecologic Surgeries During Trendelenburg Position.
Brief Title: Optic Nerve Sheath Diameter in Laparoscopic Surgeries During Trendelenburg Position
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Other Study IDs: Medipol Hospital 14
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Colon Disease; Gynecologic Disease
Keywords: Trendelenburg position; Optic nerve sheath diameter; Colon surgery; Gynecologic surgery
MeSH Terms: conditions — Colonic Diseases; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Optic nerve sheath diameter — Pre and post-trendelenburg optic nerve sheath diameter will be measured

SUMMARY:
It is difficult to measure the several levels of intracranial pressure during abdominal surgery, and direct monitoring with intracranial devices is often impossible. Measurement of optic nerve sheath diameter (ONSD) via ultrasonography has been developed as an alternative method for evaluating intracranial pressure. Increased intracranial pressure may cause in expanding of the optic nerve sheath and may increase the diameter. Therefore, measuring the diameter of the optic nerve sheath via ultrasonography is considered as a non-invasive, easy-to-apply and reliable method to evaluate intracranial pressure.

DETAILED DESCRIPTION:
The peritoneum is inflated with carbon dioxide (insufflation) and head-down position is performed (Trendelenburg) during laparoscopic colon and gynecologic surgeries. Intracranial pressure (ICP) may be affected by positive intraabdominal pressure due to pneumoperitoneum. The Trendelenburg position (usually at a degree of 25-400) causes increasing in the pressure of cerebrospinal fluid during surgery. Therefore, cerebral edema and an increasing in ICP may occur. It is difficult to measure the several levels of intracranial pressure during abdominal surgery, and direct monitoring with intracranial devices is often impossible. Measurement of optic nerve sheath diameter (ONSD) via ultrasonography has been developed as an alternative method for evaluating intracranial pressure. The optic nerve is an extension of the central nervous system, surrounded by cerebrospinal fluid (CSF) and continues with the nerve sheath. Increased intracranial pressure may cause in expanding of the optic nerve sheath and may increase the diameter. Therefore, measuring the diameter of the optic nerve sheath via ultrasonography is considered as a non-invasive, easy-to-apply and reliable method to evaluate intracranial pressure.

In this study, we aimed to evaluate the changes of optic nerve sheath diameter in patients who will undergo laparoscopic colon and gynecologic surgery during trendelenburg position. Our primary goal is to compare the optic nerve sheath diameters via ultrasonography, and our secondary aim is to evaluate the effect of this change on intracranial pressure.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for laparoscopic colon and gynecologic surgeries under general anesthesia

Exclusion Criteria:

* use of beta blocker or diuretic drugs
* severe heart failure
* diabetes with ocular or neurologic complications
* history of cardiac, eye, intracranial, and thoracic surgery
* history of hydrocephalus, glocoma, intracranial tumor, cerebrovascular disease

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Laparoscopic colon and gynecologic surgery patients aged between 18-75 years with ASA I and ASA II status will be included in this randomized prospective study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | Change from baseline optic nerve sheath diameter at 10 mins and 60 mins after trendelenburg. And 10 minutes after the re-neutral position
  Pre and post-trendelenburg diameters of optic nerve sheath

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD data

REFERENCES:
- [Background] Robba C, Cardim D, Donnelly J, Bertuccio A, Bacigaluppi S, Bragazzi N, Cabella B, Liu X, Matta B, Lattuada M, Czosnyka M. Effects of pneumoperitoneum and Trendelenburg position on intracranial pressure assessed using different non-invasive methods. Br J Anaesth. 2016 Dec;117(6):783-791. doi: 10.1093/bja/aew356. PMID 27956677
- [Background] Chen K, Wang L, Wang Q, Liu X, Lu Y, Li Y, Wong GTC. Effects of pneumoperitoneum and steep Trendelenburg position on cerebral hemodynamics during robotic-assisted laparoscopic radical prostatectomy: A randomized controlled study. Medicine (Baltimore). 2019 May;98(21):e15794. doi: 10.1097/MD.0000000000015794. PMID 31124975
- [Background] Colombo R, Agarossi A, Borghi B, Ottolina D, Bergomi P, Ballone E, Minari C, Della Porta V, Menozzi E, Figini S, Fossali T, Catena E. The effect of prolonged steep head-down laparoscopy on the optical nerve sheath diameter. J Clin Monit Comput. 2020 Dec;34(6):1295-1302. doi: 10.1007/s10877-019-00418-5. Epub 2019 Nov 5. PMID 31691148